CLINICAL TRIAL: NCT06215014
Title: Sex Effects on Blood Pressure Regulation to Acute Isometric Handgrip Exercise, Following 4 Weeks of Isometric Handgrip Training
Brief Title: Sex Effects on Blood Pressure With Handgrip Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Boston (Other)
Responsible Party: Principal Investigator, Tracy Baynard, Professor and Assoc Vice Provost, Grad Edu, University of Massachusetts, Boston
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 3471
Record Dates: First submitted 2023-09-27; First posted 2024-01-22 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Blood Pressure
Keywords: exercise training; handgrip; sex effects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Handgrip training (Experimental): Participants will perform isometric handgrip training 3 days per week for a month.
  Interventions: Other: Isometric handgrip training
- Control (No Intervention): Participants will not perform isometric handgrip training for a month.

INTERVENTIONS:
Other: Isometric handgrip training — Participants will train three days per week at home for 1 month using a reliable and validated digital handgrip dynamometer (DynX, MD System, Inc., Westerville, USA) in a seated position. The isometric handgrip training protocol will consist of four sets (2 for each hand) of two-min sustained contractions starting at 30% of maximum voluntary contraction (MVC) interspersed by 1-min resting periods (a total of 12-min). All training sessions will be remotely supervised via Zoom or phone call by a research team member to ensure compliance with the exercise prescription. Before each training session, MVCs will be re-assessed over three repetitions, each separated by 30-s, to ensure an accurate exercise prescription. The highest value will be used to determine the target intensity of the session
  Arms: Handgrip training

SUMMARY:
The goal of this intervention is to compare the blood pressure response of young females and males to a single bout of static handgrip exercise before and after static handgrip training (4 weeks).

The main questions this study aims to answer are:

* Are the lowering blood pressure effects of static handgrip exercise training different between young females and males?
* Which factors explain the lowering blood pressure effects of static handgrip training and possible differences between sexes? Is it an improved blood vessel dilation? Is it a reduced stiffening of blood vessels? Is it a reduced fight or flight response resulting in a lower heart rate and blood pumped by the heart into the vessels? All the above?
* Which factors regulate blood pressure response during and immediately after a single bout of static handgrip exercise?

All participants will be asked to:

* Visit the laboratory to perform static handgrip exercise - first visit;
* Participants will be randomized (like flipping a coin) to static handgrip exercise training or to a non-exercising phase, with each phase lasting four weeks. Participants will also complete the other condition (handgrip or no handgrip) after completing the first four-week condition
* Return to the laboratory after the completion of both static handgrip training and no training to perform the static handgrip exercise of the first visit.

The investigators will compare participants' blood pressure response to a single bout static of handgrip exercise after training to their own blood pressure response to the same bout of exercise after the non-training period.

DETAILED DESCRIPTION:
Hypertension is still the leading modifiable risk factor for cardiovascular disease and a silent independent predictor of all-cause death worldwide. Projections for the US suggest that 41% of adults will develop hypertension before 2030. Thus, it is clinically relevant to optimize interventions aimed at preventing and managing hypertension.

Isometric handgrip training holds promise to mitigate the growing prevalence of hypertension in healthy adults. This form of exercise training can be performed at home, requires less time investment compared to conventional training, and requires only one piece of inexpensive equipment. Interestingly, some but not all studies suggest that isometric handgrip training yields superior antihypertensive effects in young healthy males compared to their female counterparts. The mechanisms behind the antihypertensive effects of isometric handgrip training are yet to be determined. Possible candidates include: 1) increases in cardiovagal modulation and 2) increases in endothelial nitric oxide-dependent vasodilation coupled with reductions in arterial stiffness.

The understanding of blood pressure (BP) regulation to acute isometric handgrip exercise would provide valuable mechanistic insight into possible sex-dependent antihypertensive effects of this form of training, given that acute responses likely translate into antihypertensive training adaptations. In fact, in healthy young adults, an acute bout of isometric handgrip exercise has been shown to evoke a higher blood pressure response in males compared to females immediately after exercise cessation. Given that higher hypertensive responses to acute isometric handgrip exercise are associated with greater reductions in resting BP following isometric handgrip training, this could explain the larger antihypertensive effects reported in young males. Importantly, young females are generally less fatigable to isometric handgrip exercise performed at the same relative intensity than males. This sex difference in muscle fatigability relates to the larger muscle mass and strength of males leading to higher intramuscular pressures that compress feeding arteries but also to the smaller increments in blood pressure of females to exercise. Importantly, whether this sex difference in fatigability and blood pressure during acute isometric handgrip exercise limits the potential for blood pressure-related adaptations to handgrip training in females is unknown. In addition, young females also exhibit a faster BP recovery to acute isometric handgrip exercise than their male counterparts. Mechanistically, this faster recovery is, in part, attributed to faster cardiovagal reactivation and higher increases in baroreflex sensitivity observed in females but not in males. However, whether other regulatory mechanisms, such as increases in endothelial nitric oxide-mediated vasodilation and or reductions in sympathetic outflow to blood vessels contribute to this apparently faster blood pressure recovery in females after a hypertensive stimulus is unknown. In addition, blood flow and baroreflex dynamics interplay during isometric handgrip exercise are largely unknown which might provide valuable insight into blood pressure regulation after exercise cessation.

Therefore, the specific aims of this study are threefold:

Aim 1 - To examine if the effects of a 4-week isometric handgrip training intervention on BP regulation to a fatiguing bout of isometric handgrip exercise are sex- dependent in young healthy adults with normal BP

Aim 2 - To examine if blood pressure responses are sex-dependent during and after a fatiguing bout of isometric handgrip exercise at 30% maximum voluntary contraction in healthy young adults with normal blood pressure;

Aim 3 - To determine the effects of sex on the regulatory mechanisms of blood pressure, including cardiac autonomic and vascular function during and after a fatiguing bout of isometric handgrip exercise in healthy young adults with normal BP.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 18-40 years;
* Normal blood pressure as defined by the American Heart Association (<130/90 mmHg);
* BMI < 30 kg/m2;
* No cardiovascular risk factors and no clinically diagnosed cardiovascular disease;
* Being recreationally active (≤ 2 days of structured physical activity);
* Able to speak English.

Exclusion Criteria:

* Diagnosed with cardiovascular disease (e.g., coronary artery disease, heart failure), musculoskeletal (i.e., osteoporosis and sarcopenia), metabolic disease (e.g., diabetes mellitus) and kidney disease;
* Taking antihypertensive or other vasoactive medications and cardioactive medication;
* Diagnosed with depression and/or anxiety disorders;
* Long COVID;
* Being a smoker;
* Being pregnant or having menstrual irregularities.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Brachial blood pressure | "Baseline, pre-intervention/oscillometry", "Within 5-days after the intervention/oscillometry"
  Systolic and diastolic blood pressure
Flow-mediated dilation | "Baseline, pre-intervention/ultrasonography", "Within 5-days after the intervention/ultrasonography"
  Non-invasive measurement of endothelial function
Root mean square of successive differences (RMSSD) | "Baseline, pre-intervention/electrocardiography", "Within 5-days after the intervention/electrocardiography"
  Heart rate variability metric of the time domain reflecting cardiovagal modulation
High frequency power band | "Baseline, pre-intervention/electrocardiography", "Within 5-days after the intervention/electrocardiography"
  Heart rate variability metric of the spectral domain reflecting cardiovagal modulation
Carotid femoral pulse wave velocity (cfPWV) | "Baseline, pre-intervention/ultrasonography", "Within 5-days after the intervention/applanation tonometry"
  Central arterial stiffness

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Baynard, PhD, Principal Investigator — University of Massachusetts, Boston
Locations (2):
- United States (2):
  - UMassachusetts Boston, Boston, Massachusetts
  - University of Massachusetts Boston, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-19): https://cdn.clinicaltrials.gov/large-docs/14/NCT06215014/Prot_SAP_000.pdf
  • Informed Consent Form (2023-10-19): https://cdn.clinicaltrials.gov/large-docs/14/NCT06215014/ICF_001.pdf